CLINICAL TRIAL: NCT05423587
Title: Genicular artEry embolisatioN in patiEnts With oSteoarthrItiS of the Knee II
Brief Title: Genicular Artery Embolisation for Knee Osteoarthritis II
Acronym: GENESISII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VAR-2021-11; 286849 (Other: IRAS)
Record Dates: First submitted 2022-04-11; First posted 2022-06-21 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Knee Osteoarthritis
Keywords: Microspheres; Embozene; Artery Embolization; Joint diseases; Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases

STUDY DESIGN:
Intervention Model Description: Single Site, Double Blind Sham Randomized Controlled Trial with Sham subject optional crossover to the treatment arm (GAE) at 6 months post randomization to determine if embolization of abnormal blood vessels arising from branches of the genicular arteries reduces pain in patients with knee osteoarthritis.
Who Masked: Participant, Care Provider
Masking Description: A randomization algorithm (hidden and protected) allocates a random number to each of the 110 subjects. The outputs of this algorithm will only be accessible to those who are unrestricted by experimental blinding (operator, radiographer, scrub nurse). For safety reasons the interventional radiologist will be aware of the treatment arm (non-blind).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GAE Treatment (Experimental): The genicular artery embolisation procedure identifies abnormal blood vessels in the knee via angiogram imaging. Through groin access and puncture of the femoral artery through a small sheath tiny microspheres (Embozene(TM)) will be injected into this area and reduce blood flow in order to reduce pain.
  Interventions: Procedure: Genicular Artery Embolisation
- Sham Procedure (Sham Comparator): In the control (sham) arm patients will not undergo the embolisation procedure with microspheres, instead they will have 2ml of saline injected into their knee artery supplying the abnormal area of the knee. The remainder of the procedure is otherwise identical between the two groups.
  Interventions: Procedure: Genicular Artery Injection

INTERVENTIONS:
Procedure: Genicular Artery Embolisation — Transarterial catheter directed embolisation of hypervascularity in patients with mild to moderate knee osteoarthritis
  Other Names: Embozene Microspheres; Embozene
  Arms: GAE Treatment
Procedure: Genicular Artery Injection — Transarterial catheter directed injection of normal (0.9%) saline in patients with mild to moderate knee osteoarthritis
  Arms: Sham Procedure

SUMMARY:
This clinical study is designed as a double-blind sham controlled randomised trial with the option of sham group crossover to receive the GAE treatment at 6 months after unblinding. This study will determine if embolisation of abnormal neovasculature arising from branches of the genicular arteries reduces pain in patients with knee osteoarthritis. The study patient population will consist of up to 110 subjects with knee pain for at least 3 months that is resistant to conservative treatment measures. Subjects will be treated with knee embolisation or 2 mL of saline in the sham arm. At 6 months, all subjects in the sham arm will be allowed to cross-over and receive the embolisation procedure with a follow-up duration of 18 months. The total planned study duration is 3.5 years.

DETAILED DESCRIPTION:
This is a single-center, randomised trial to compare patients who receive genicular artery embolisation of the knee with patients who receive a sham procedure with saline injection.

The study population will consist of up to 110 subjects with knee pain that is resistant to conservative treatment measures for at least 3 months. Subjects will be followed for 24 months. At 6 months patients will be unblinded and offered an optional crossover to receive the GAE procedure with 18 months follow-up.

Alongside a sham surgery placebo arm, a high-quality systematic review of surgical RCTs was used as a suitable benchmark to inform the sample size and power calculation.

With a 0-100 scale for the primary endpoint of KOOS4, assuming a 1:1 randomization, a mean difference of 6.4 (i.e., effect size) between GAE and Sham treatments, a common standard deviation of 10 (i.e., a Cohen's D of 0.64), an alpha error of 2-sided 0.05 and a power of 0.85, the 2-arm total sample size the requirement is 88 subjects (44 each arm) by Normal approximation. Allowing for a participant dropout rate of 20%, the enrolment goal is 110 participants, approximately 55 in each study arm.

All study subjects will undergo a physical exam and history, a contrast-enhanced knee MRI, blood serum and neuropschological assessment with a functional head MRI to identify potential predictors of treatment success.

In the GAE treatment arm subject will undergo a genicular artery embolization with Embozene microspheres (100 micron) (Varian Medical Systems) and the Sham group will receive saline through the transarterial catheter through groin access.

Participants will be randomly assigned to have particulate embolisation with 100-micron Embozene particles, or to injection with 2 ml heparinized normal saline (sham arm) At 6 months participants will be unblinded and there will be an open extension period for 6 months, in which participants in the sham arm will be offered GAE.

Follow-up visits will be at 1 month, 3 months, 6 months, 12 months and 24 months post randomisation. At these visits subjects will complete the KOOS score, the visual analog scale (VAS) pain score, an analgesia diary, and at specific time points the EQ-5D-3L, and report any new adverse events (AEs).All subjects will undergo a contrast-enhanced knee MRI at baseline and at 6 and 12 months.

At 6 months after unblinding the sham group subjects have the option to cross over and receive the GAE treatment with follow-up at 1 month, 3 months, 6 months, 12 months and 18 months.

ELIGIBILITY:
Inclusion Criteria:

ALL inclusion criteria below need to be fulfilled for the patient to participate in the study.

* Participant is willing and able to give informed consent for participation in the study.
* Participants aged 45 years or above.
* Grade 1-3 knee OA on X-ray as per Kellgren-Lawrence Grading Scale
* Knee pain for at least 3 months resistant to conservative non-surgical treatment (e.g., physiotherapy, steroid injections, weight loss programs, PRP (platelet-rich plasma) injections)
* Be able to lie flat for at least 6 hours-this will be assessed by asking how participants sleep (bed, chair recumbent, semi-recumbent) and assessing what prevents them from lying flat overnight (breathlessness, back pain, etc)
* Minimum score of 50 on baseline 0 - 100 VAS

Exclusion Criteria:

The patient may not enter the study if ANY of the following apply:

* Rheumatoid arthritis or infectious arthritis
* Severe knee OA (grade 4 on x-ray as per Kellgren-Lawrence Grade)
* Renal impairment: eGFR <45. Assessed from medical records or a blood test if required as is part of standard clinical practice when considering a patient for a therapeutic intervention.
* Patients with a bleeding diathesis, or other bleeding risk such as patients on warfarin which cannot be stopped easily (e.g., patients with metallic heart valves) assessed by asking the patient and from medical records. Uncorrectable bleeding diathesis: INR>1.6, Platelets <50,000
* Requires oxygen on ambulation. Assessed by asking the patient and from medical records.
* Low life expectancy (<1 year)
* Communication difficulty due to language barriers
* Contraindication to MRI
* Known allergies to barium sulfate, 3-aminopropyltrialkoxysilane, polyphosphazene or IV radiopaque contrast agent
* History of Peripheral Arterial Disease (PAD) with intermittent claudication and/or rest pain
* Pregnancy or positive pregnancy test (the participant will be exposed to ionising radiation during the fluoroscopy procedure)
* Any other significant disease or disorder which, in the opinion of the recruiting physician, may put the participants at risk because of participation in the study, or may influence the result of the study or the participant's ability to participate

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-10-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Determine if embolisation of abnormal neovasculature arising from branches of the genicular arteries reduces pain in patients with knee OA compared to Sham treatment | 6 months
  Change from baseline to 6 months post randomisation in the mean score on four Knee Injury and Osteoarthritis Outcome Score subscales, covering pain, symptoms, activities of daily living, and quality of life (KOOS4); scores range from 0 (worst) to 100 (best)

SECONDARY OUTCOMES:
Determine clinical success | 6 months
  The proportion of subjects reporting at least a 10- point improvement in KOOS scores at 6-months (where a 10-point change from baseline is defined as the minimum clinically important difference (MCID)
Assessment of pain relief | 6 months
  Pain relief at 6 months post randomisation, using the patient-reported 0 - 100 visual analogue scale (VAS) pain score
Determine if embolisation improves pain, function, and quality of life in patients with knee OA compared to Sham treatment | 6 months
  All 5 subscales of the KOOS questionnaire will be analysed at 6 months post randomisation.

OTHER OUTCOMES:
Determine safety and toxicity | 6 months follow-up
  Proportion of subjects experiencing relevant adverse events (as per SIR Adverse Event Classification System) at 6 months post randomisation
Determine if improvement of knee osteoarthritis can be described by imaging analysis following GAE vs Sham | 6 months
  Whole Organ Magnetic Resonance Imaging Score (WORMS) for non-invasive assessment of synovial hypertrophy and neo-vascularization for osteoarthritis at 6 months post randomisation.
Quantification of a personalised psychometric pain profile to determine whether treatment response can be predicted using behavioural indicators of predisposition to central facilitation of pain | 6 months
  Pain Catastrophizing Scale (PCS) patient questionnaire: Score reflects on painful experiences of the patient. Score from 0 (minimum) to 52 (maximum). A higher score means worse outcome
Determine quality of life changes | 6 months
  Changes in quality of life measured by Euro-Quality of Life-5D-3L (EQ-5D-3L) assessing five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), each having three levels (3L): no problems, some problems, extreme problems (labelled 1-3) in a descriptive fashion.
Assess patient reported acceptability of study treatment | 1 week after treatment
  The PROM questionnaire (Patient reported outcome measures) (10 question patient questionnaire) reports scores between 9 (minimum) to 90 (maximum) where a high score is considered worse acceptance (worse outcome)
Determine if patient's need for analgesia will be reduced | 6 months
  Change of analgesia intake at 6 months post randomisation.
Assess durability of GAE | 24 months
  Time to failure, i.e., time to next invasive intervention for those receiving GAE treatment following (a) randomisation, or (b) crossing over to GAE from Sham arm.
Perform a health economic cost effectiveness analysis of GAE versus other treatment modalities in the moderate knee OA space | 6 months
  Changes in quality of life measured by EuroQoL-5D (EQ-5D-3L) combined with the time assessment to failure (durability of GAE), i.e., time to next invasive intervention for those receiving GAE treatment following (a) randomization, or (b) crossing over to GAE from Sham arm will be assessed together to describe the cost effectiveness.
Determine if embolisation improves pain, function, and quality of life in patients with knee OA in the treatment group | 24 months follow-up
  All 5 subscales of the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire will be analysed at 12 and 24 months post randomisation. Scores range from 0 (minimum, worst) to 100 (maximum, best).
Determine quality of life changes in the GAE group at 12 and 24 months | 24 months follow-up
  Changes in quality of life measured by Euro-Quality of Life-5D-3L (EQ-5D-3L) assessing five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression, each having three levels (3L): no problems, some problems, extreme problems (labelled 1-3) at 12 and 24 months post randomisation in a descriptive fashion.
Describe imaging outcomes of knee at 12 months in GAE | 12 months
  Whole Organ Magnetic Resonance Imaging Score (WORMS) for non-invasive assessment of synovial hypertrophy and neo-vascularization for osteoarthritis will be evaluated in the GAE group at 12 months post randomisation.
Determine if patient's need for analgesia will be reduced in the GAE group | 24 months
  Change of analgesia intake at 12 and 24 months post randomisation.
Assessment of pain relief in the GAE group | 24 months
  Pain relief at 12 and 24 months post randomisation, using the patient-reported 0 - 100 visual analogue scale (VAS) pain score
Determine if embolisation improves pain, function, and quality of life in patients with knee OA in the treatment group and compare with the Sham group in subjects who do not cross over at 12 and 24 months | 24 Months
  All 5 subscales of the Knee Injury and Osteoarthritis Outcome Score (KOOS) will be analysed at 12 and 24 months post randomisation in the GAE and Sham group. Scores range from 0 (worst) to 100 (best).
Determine quality of life changes in the GAE and sham group | 24 months
  The second part of the Euro-Quality of Life-5D-3L questionnaire consists of a visual analytic scale (VAS) on which the patient rates his / her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health) at 12 and 24 months post randomisation in the GAE group and compare with the Sham group in subjects who do not cross over.
Determine if patient's need for analgesia will be reduced | 24 months
  Compare changes of analgesia intake at 12 and 24 months post randomisation in the GAE group with the Sham group in subjects who do not cross over.
Assessment of pain relief | 24 months
  Compare pain relief in the GAE group at 12 and 24 months post randomisation, using the patient-reported 0 - 100 visual analogue scale (VAS) pain score, and compare to the Sham group in subjects who do not cross over.
Determine if embolisation improves pain, function, and quality of life in patients with knee OA in the Sham crossover group at 1, 3, 6, 12 and 18 months | 18 months
  All 5 subscales of the Knee Injury and Osteoarthritis Outcome Score (KOOS) will be analysed at 1,3,6, 12 and 18 months post treatment in the Sham crossover group. Scores range from 0 (worst) to 100 (best).
Assessment of pain relief in the Sham crossover group | 18 months
  Pain relief at 1,3,6,12 and 18 months post treatment in the Sham crossover group, using the patient-reported 0 - 100 visual analogue scale (VAS) pain score
Determine if patient's need for analgesia will be reduced in the Sham crossover group | 18 months
  Change of analgesia intake at 1,3,6,12 and 18 months post treatment in the Sham crossover group.
Determine quality of life changes in the Sham crossover group | 18 months
  Changes in quality of life measured by Euro-Quality of Life-5D-3L (EQ-5D-3L) assessing five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression, each having three levels (3L): no problems, some problems, extreme problems (labelled 1-3) at 6, 12 and 18 months post treatment in a descriptive fashion.
Determine if improvement of knee osteoarthritis can be described by imaging analysis in the Sham crossover group following GAE | 12 months
  Whole Organ Magnetic Resonance Imaging Score (WORMS) for non-invasive assessment of synovial hypertrophy and neo-vascularization for osteoarthritis at 6 and 12 months post treatment in the Sham crossover group
Quantification of mindfulness as part of a personalised psychometric pain profile to determine whether treatment response can be predicted using behavioural indicators of predisposition to central facilitation of pain | 6 months
  Five-Facet Mindfulness Patient Questionnaire (FFMQ): Reporting a score between 15 (minimum) and 75 (maximum). Higher scores are better and indicative of high trait mindfulness.
Assessment of depressive symptoms as part of a personalised psychometric profile | 6 months
  Patient Health Questionnaire (PHQ-9): Reports a score between 0 (minimum) and 27 (maximum) with higher scores being worse representing high depressive symptoms
Assessment of patient's psychological flexibility as part of personalised psychometric profile | 6 months
  Pain Interference - Short Form 6b (PROMIS) patient questionnaire: Reports a score between 6 (minimum) and 30 (maximum), with higher scores being worse representing high pain interference
Assessment of a patient's anxiety as part of a personalised psychometric profile | 6 months
  Generalized Anxiety Disorder (GAD-7) patient questionnaire: reports a score between 0 (minimum) and 21 (maximum). Higher scores are worse representing more severe levels of anxiety.
Quantification of patient's psychological flexibility as part of a personalised psychometric profile | 6 months
  Committed Action Questionnaire (CAQ-8): Reports a score between 0 (minimum) and 48 (maximum). Higher scores mean better outcome representing high commitment to goals.
Quantification of a patient's intolerance of uncertainty | 6 months
  Intolerance of Uncertainty Scale - Short Form patient questionnaire: Reports a score between 0 (minimum) and 60 (maximum). Higher scores are worse representing high intolerance of uncertainty.
Quantification of a patient's sleep quality as part of personalised psychometric profile | 6 months
  Pittsburgh Sleep Quality Index (PSQI) patient questionnaire: Reports a score between 0 (minimum) to 21 (maximum). Higher scores are worse indicating worse sleep quality.
Assessment of psychological inflexibility in pain as part of a personalised psychometric pain profile to determine whether treatment response can be predicted using behavioural indicators of predisposition to central facilitation of pain | 6 months
  Psychological Inflexibility in Pain Scale (PIPS) patient questionnaire: reports scores between 16 (minimum) to 112 (maximum). Higher scores (worse results) indicate low flexibility in regard to dealing with pain.
Quantification of the perspective of a participant's viewpoint on pain as part of a personalised psychometric pain profile | 6 months
  Pain Priors Questionnaire
Behavioural quantification of psychological flexibility to stratify patients who achieve optimal clinical outcomes from the treatment procedure. | 6 months
  Wisconsin Card Sorting Task: reports reaction time measured in milliseconds (lower value is better outcome as better cognitive function)
Assess functional connectivity between brain regions and investigate the influence of metabolite levels within pain modulatory regions as a neurochemical marker for vulnerability to further chronic pain states. | 6 months
  Functional head MRI
Assess patient's capacity of central pain modulation | 6 months
  Quantitative sensory testing: Central pain modulation (CPM) measures the degree to which pain at one site inhibits pain at a distal site. The difference between the initial and final rating is taken as a score of the participant's CPM capacity with a range of -10 to 10 with -10 representing a better result with high pain inhibition/modulation.
Assess patient's intrinsic attention to pain | 6 months
  Intrinsic Attention to Pain (IAP) test measures whether a participant's attention is intrinsically gravitated towards, or away from pain during thermal stimulation with a score range of +2 to -2, with + 2 representing worse results indicating an inability to attentionally disengage from pain.
Assess patient's capacity of central facilitation of pain | 6 months
  Temporal Summation (TS) test: describes the degree to which pain responses are centrally enhanced by rapid repeated presentation. A score between -10 to 10 is reported with 10 representing high pain summation as a worse result and -10 no pain summation.
Perception of health by patient in the GAE and sham group | 6 months
  The second part of the Euro-Quality of Life-5D-3L questionnaire consists of a visual analytic scale (VAS) on which the patient rates his / her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).
Perception of health by patient in the GAE group | 24 months follow-up
  The second part of the Euro-Quality of Life-5D-3L questionnaire consists of a visual analytic scale (VAS) on which the patient rates his / her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).
Perception of health by patient in GAE and sham group at 12 and 24 months | 24 months
  The second part of the Euro-Quality of Life-5D-3L questionnaire consists of a visual analytic scale (VAS) on which the patient rates his / her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health) at 12 and 24 months post randomisation in the GAE group and compare with the Sham group in subjects who do not cross over.
Perception of health by patient in sham crossover group at 6, 12 and 18 months | 18 months
  The second part of the Euro-Quality of Life-5D-3L questionnaire consists of a visual analytic scale (VAS) on which the patient rates his / her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health) at 6, 12 and 18 months post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Little, MD, Principal Investigator — Royal Berkshire NHS Foundation Trust, Reading, UK
Locations (1):
- Royal Berkshire NHS Foundation Trust, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Little MW, Harrison R, MacGill S, Speirs A, Briggs JH, Tayton E, Davies NLC, Hausen HS, McCann C, Levine LL, Sharma RA, Gibson M. Genicular Artery Embolisation in Patients with Osteoarthritis of the Knee (GENESIS 2): Protocol for a Double-Blind Randomised Sham-Controlled Trial. Cardiovasc Intervent Radiol. 2023 Sep;46(9):1276-1282. doi: 10.1007/s00270-023-03477-z. Epub 2023 Jun 19. PMID 37337060